CLINICAL TRIAL: NCT03947307
Title: Kinesiotape Treatment for Postoperative Edema After Joint Replacement Surgery of the Knee -The KNEETAPE Study
Brief Title: Kinesiotape Treatment for Postoperative Edema After Joint Replacement Surgery of the Knee- The KNEETAPE Study
Acronym: KNEETAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-00219; ch19Saxer3
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Edema
Keywords: total knee replacement; Kinesiotape treatment; manual lymphatic drainage; compressive bandages; Kinesiotaping

STUDY DESIGN:
Intervention Model Description: comparing the use of kinesiotape for the treatment of postoperative edema after knee joint arthroplasty to standard treatment (manual lymphatic drainage and compression in form of stockings or compressive bandages), as well as to sham interventional treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blind to the difference between kinesio- and sham-taping, allowing a double blinded design for the evaluation of the effect of kinesio- versus other tapes. Patient blinding for kinesiotaping versus manual lymphatic drainage is not feasible. The assessment of the primary outcome i.e. the assessment of leg circumference on day 1 and 8 will be performed by a blinded assessor unaware of the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Intervention (treatment / medical device) (Experimental): Patients in the experimental group will receive lymphtaping using Easytape® according to common practice on day 1 after surgery by specifically trained physiotherapists. The tape has an elasticity of 150%. The material is moisture- and air-permeable with a hypoallergenic adhesive coating that is activated by body temperature to increase durability of contact. If possible the taping will be left for 7 days, in case of insufficient adhesion taping will be repeated.
  Interventions: Device: lymphtaping using Easytape®
- Control Intervention (compression treatment ) (Active Comparator): Patients in the control group will be treated with manual lymphatic drainage followed by compression treatment using compressive stockings if accepted or compressive bandaging in cases with pronounced swelling depending on medical necessity.
  Interventions: Procedure: compression treatment
- Control Intervention (sham taping) (Sham Comparator): Patients in the control group will be treated by sham taping with Leukotape® Classic, a non-elastic tape, that in all other respects resembles Easytape®.
  Interventions: Device: sham taping

INTERVENTIONS:
Device: lymphtaping using Easytape® — lymphtaping using Easytape® on day 1 after surgery by specifically trained physiotherapists. If possible the taping will be left for 7 days.
  Arms: Experimental Intervention (treatment / medical device)
Procedure: compression treatment — manual lymphatic drainage followed by compression treatment using compressive stockings or compressive bandaging
  Arms: Control Intervention (compression treatment )
Device: sham taping — sham taping with Leukotape® Classic, a non-elastic tape, that in all other respects resembles Easytape®.
  Arms: Control Intervention (sham taping)

SUMMARY:
Postoperative edema is a common condition affecting wound healing and function. Traditionally, manual lymphatic drainage and compressive bandages have been employed to reduce swelling. Kinesiotaping might be an alternative approach. To analyse the efficacy, cost-effectiveness, satisfaction, quality of life, functional outcome and and morbidity of the use of kinesiotape for the treatment of postoperative edema after knee replacement surgery, compared to standard manual lymphatic drainage with compression (i.e. compressive stockings or bandages) or sham taping.

ELIGIBILITY:
Inclusion Criteria:

* Joint replacement surgery of the knee including conversion from partial to total joint replacement or revision surgery
* Informed Consent as documented by signature

Exclusion Criteria:

* Isolated retropatellar replacement or revision surgery for infection
* Contraindications to manual lymphatic drainage and compression treatment (i.e. compressive stockings or bandages) e.g. heart failure
* Contraindication to kinesiotape treatment, e.g. hypersensitivity to medical glue
* Dermatoses at or around the surgical site
* Suspected or confirmed local infection
* Participation in another trial with investigational drug within the 30 days preceding and during the present trial
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Inability for consent or assent by the patient, or lack of proxy consent in assenting patients with signs of incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Change in leg circumference between day 1 and day 8 (in cm) | day 1 postoperatively before start of intervention and every day thereafter for 7 days
  Leg circumference will be measured at three levels (joint space, 5cm proximal, 5cm distal) with each three measurements performed by one assessor in all patients and time points. The primary endpoint will be the mean of the three measurements

SECONDARY OUTCOMES:
Change in leg circumference between day 0 and day 8 (in cm) | day 0 preoperative and day 1 postoperatively before start of intervention and every day thereafter for 7 days
  Leg circumference will be measured at three levels (joint space, 5cm proximal, 5cm distal) with each three measurements performed by one assessor in all patients and time points. The primary endpoint will be the mean of the three measurements
Change in leg circumference between day 0 and after 6 weeks and 12 weeks (in cm) | day 0 preoperative and after 6 weeks and 12 weeks after start of intervention
  Leg circumference will be measured at three levels (joint space, 5cm proximal, 5cm distal) with each three measurements performed by one assessor in all patients and time points. The primary endpoint will be the mean of the three measurements
Change in range of motion of knee (in degree) | day 1 postoperatively before start of intervention and at day 8 after start of intervention and after 6 and 12 weeks after start of intervention
  range of motion measured using the neutral zero method

OTHER OUTCOMES:
Change in Quality of life assessment (EQ5D-5L) | assessed on day 0 preoperative, day 8 and week 12 after start of intervention
  assessment of 5 dimensions of life: mobility, self-care, activities of daily living, pain and psychological well-being in each 5 categories ranging from "no problems" to "extreme problems"
Change in patient satisfaction with the received treatment (VAS) | assessed on day 8 and week 12 after start of intervention
  visual analogous scale (VAS) on which the patient can rate satisfaction with the received treatment; Scale from 0 = not at all satisfied to10 = very satisfied
Change in Knee disability and Osteoarthritis Outcome Score (KOOS) | assessed on day 8 and week 12 after start of intervention
  Patient reported score. The KOOS results in summary scores for five subscales. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec) and knee-related Quality of Life (QOL). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee Problems.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Egloff, Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Department of Orthopaedics and Trauma Surgery (DOTS)., Basel, Switzerland